CLINICAL TRIAL: NCT04044417
Title: Curcumin-Simvastatin Release Profile in the Gingival Crevicular Fluid Following EDTA Root Surface Etching in the Surgical Treatment of Intrabony Periodontal Defects - A Biochemical and Clinical Study
Brief Title: Curcumin-Simvastatin-EDTA in the Treatment of Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Eman Farouk Mohamed Hussein Elsobky, demonstrator of oral medicine and periodontology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FER16 21-M
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Periodontitis
Keywords: periodontitis; curcumin; simvastatin; EDTA
MeSH Terms: conditions — Periodontitis | interventions — Curcumin; Simvastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- open flap debridement only (Placebo Comparator): surgical treatment of periodontal defects
  Interventions: Procedure: currettage
- curcumin and simvastatin (Active Comparator): open flap debridement followed by application of curcumin-simvastatin paste (2% curcumin and 1.2% simvastatin).
  Interventions: Procedure: currettage; Drug: curcumin simvastatin paste
- EDTA, curcumin and simvastatin (Active Comparator): open flap debridement followed by 24% EDTA root surface etching and application of curcumin-simvastatin paste (2% curcumin and 1.2% simvastatin).
  Interventions: Procedure: currettage; Drug: curcumin simvastatin paste; Drug: EDTA root conditioning

INTERVENTIONS:
Procedure: currettage — open flap debridement
  Other Names: surgical treatment of periodontal defects
Drug: curcumin simvastatin paste — Curcumin is the primary active constituent of turmeric. Simvastatin is chemical modification of lovastatin.
  Other Names: open flap debridement followed by application of curcumin-simvastatin paste (2% curcumin and 1.2% simvastatin).
  Arms: EDTA, curcumin and simvastatin; curcumin and simvastatin
Drug: EDTA root conditioning — EDTA is an aminopolycarboxylic acid and a colourless, water-soluble solid
  Other Names: open flap debridement followed by 24% EDTA root surface etching and application of curcumin-simvastatin paste (2% curcumin and 1.2% simvastatin).
  Arms: EDTA, curcumin and simvastatin

SUMMARY:
Among the root conditioning materials is the Ethylenediaminetetraacetic acid (EDTA). EDTA exposes the collagen fibers on dentin surfaces and also enhances early cell colonization. Statins have an anti-inflammatory effect, inhibit the bone resorption and stimulate the bone formation. Curcumin is effective in preventing periodontal disease destruction by targeting both bacteria and host inflammatory cells. Curcumin has anti- inflammatory, antioxidant, anticarcinogenic, antiviral, and antimicrobial functions. This study will be carried out to examine the effect of simvastatin-curcumin paste following EDTA root surface etching when used in conjunction with open flap debridement treating deep periodontal pockets (suggesting that it may have positive effect)

DETAILED DESCRIPTION:
The present study entailed thirty patients having stage II or stage III, Grade A periodontitis with 30 intrabony defects. Patients were divided into three groups; group I was subjected to open flap debridement only. Group II was subjected to open flap debridement followed by application of curcumin-simvastatin paste (2% curcumin and 1.2% simvastatin). Group III was subjected to open flap debridement followed by 24% EDTA root surface etching and application of curcumin-simvastatin paste (2% curcumin and 1.2% simvastatin).Clinical parameters including plaque index, sulcus bleeding index, probing depth and clinical attachment level were recorded pre-surgical. Moreover, radiographic examination was performed by cone beam computed tomography (CBCT) just before the surgery . Vertical bone defects were exposed by full thickness mucoperiosteal flap following intrasulcular incision and thorough debridement was performed. Group II received local application of curcumin-simvastatin paste .Group III received curcumin-simvastatin paste after debridement and 24 % EDTA. The same initial clinical parameters were recorded three and six months postoperatively. Radiographic measurements were recorded six months post surgically.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering at least a single posterior 2-3 wall periodontal Pocket of depth ≥ 5 mm, attachment loss ≥3 mm, intrabony component ≥3 mm, plaque index ≤1 (Sillness and Loe, 1964) and sulcus bleeding index ≤1 (Mühlemann & Son, 1971). All these criteria were determined after phase I conventional periodontal therapy.
* Systemically healthy as evidenced by burket's oral medicine health history question questionnaire (Glick et al., 2008).
* Patients available during follow-up periods

Exclusion Criteria:

* Smoking
* Patient unwilling to comply with periodontal hygienic instructions
* Patients under any long-term chronic medication
* Vulnerable individuals

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08-25 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2018-10-03 (Actual)

PRIMARY OUTCOMES:
clinical score | change from base line to 6 months
  Probing depth (PD): evaluate the average reduction in probing depth measured in millimeters. Reduction in probing depth indicates that EDTA, simvastatin, and curcumin have positive effects in treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Y Gamal, Professor, Study Director — Faculty of dentistry- Ain shams university

IPD SHARING:
Plan to Share IPD: No